CLINICAL TRIAL: NCT01975116
Title: A Phase I Trial of p28 (NSC745104), a Non-HDM2 Mediated Peptide Inhibitor of p53 Ubiquitination in Pediatric Patients With Recurrent or Progressive CNS Tumors
Brief Title: p28 in Treating Younger Patients With Recurrent or Progressive Central Nervous System Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-041; NCI-2013-01710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-041 (Other: Pediatric Brain Tumor Consortium); PBTC-041 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Teratoid Tumor, Atypical; Choroid Plexus Neoplasms; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Brainstem Tumors; Giant Cell Glioblastoma; Glioblastoma; Gliosarcoma; Medulloblastoma; Neuroectodermal Tumor, Primitive
MeSH Terms: conditions — Teratoid Tumor, Atypical; Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Brain Stem Neoplasms; Glioblastoma; Gliosarcoma; Medulloblastoma; Neuroectodermal Tumors, Primitive | interventions — azurin (50-77)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment: p28 (Experimental): Pts receive azurin-derived cell-penetrating peptide p28 IV over 15 min 3x/week for 4 wks. Tx repeats every 6 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: azurin-derived cell-penetrating peptide p28

INTERVENTIONS:
Drug: azurin-derived cell-penetrating peptide p28 — Given IV
  Other Names: azurin-derived CPP p28

SUMMARY:
This phase I trial studies the side effects and best dose of azurin-derived cell-penetrating peptide p28 (p28) in treating patients with recurrent or progressive central nervous system tumors. Drugs used in chemotherapy, such as azurin-derived cell-penetrating peptide p28, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish whether the adult recommended phase II dose of 3x/week bolus infusions of p28is safe for pediatric patients with recurrent/refractory central nervous system (CNS) tumors.

II. To describe dose-limiting toxicities of 3x/week bolus infusions of p28 in pediatric patients with recurrent/refractory CNS tumors.

III. To evaluate and characterize the plasma pharmacokinetics of p28 in children with recurrent/ refractory CNS tumors.

SECONDARY OBJECTIVES:

I. To describe in the context of a phase I trial any observed antitumor activity of p28.

II. To investigate levels of p53 in clinical tumor specimens of patients with pediatric gliomas and other pediatric CNS tumors treated with p28.

III. To document the type/site(s) of p53 mutation in tumor tissue specimens. IV. To evaluate and characterize the intratumoral pharmacokinetics of p28 in children with recurrent/ refractory CNS tumors, if available.

OUTLINE: This is a dose-escalation study.

Patients receive azurin-derived cell-penetrating peptide p28 intravenously (IV) over 15 minutes thrice weekly for 4 weeks. Treatment repeats every 6 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed primary progressive, recurrent or refractory CNS tumors with no known curative therapies limited to high grade glioma, such as glioblastoma multiforme, medulloblastoma, primitive neuroectodermal tumor, atypical teratoid/rhabdoid tumor, anaplastic astrocytoma, high-grade astrocytoma not otherwise specified (NOS), anaplastic oligodendroglioma, or choroid plexus carcinoma; or diffuse intrinsic pontine glioma; the requirements for histological verification are waived for diffuse intrinsic pontine glioma
* Patients must not have received myelosuppressive chemotherapy or immunotherapy within 3 weeks of registration (6 weeks if prior nitrosourea)
* Patients must have received their last dose of biologic agent >= 7 days prior to study registration
* Steroid dose should be stable or decreasing for at least 1 week prior to registration
* If prior therapy was monoclonal antibody, 30 days or 3 half-lives must have elapsed (whichever is longer), prior to registration
* Patient must be off all colony stimulating factors > 1 week prior to registration (filgrastim [GCSF], sargramostim [GM CSF], erythropoietin)
* Any craniospinal irradiation must have taken place >= 3 months prior to registration >= 8 weeks for local irradiation to primary tumor; >= 2 weeks prior to study entry for focal irradiation for symptomatic metastatic sites
* Karnofsky performance scale (KPS) (for > 16 years [yrs] of age) or Lansky performance score (LPS) (for =< 16 years of age) >= 50 assessed within two weeks prior to registration
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to registration
* Absolute neutrophil count >= 1000/ mm^3 (unsupported)
* Platelets >= 100,000/ mm^3 (unsupported)
* Hemoglobin >= 8g/dL (with or without packed red blood cells [PRBC] transfusion)
* Total bilirubin =< 1.5 times upper limit of normal for age
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 times institutional upper limit of normal for age
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3.0 times institutional upper limit of normal for age
* Blood glucose within normal limits for age (If above institutional normal limits must be repeated as fasting and then within normal limits [WNL] for age)
* Creatinine clearance or nuclear glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age as follows:

  * =< 5 years: 0.8 mg/dL
  * > 5 to =< 10 years: 1 mg/dL
  * > 10 to =< 15 years: 1.2 mg/dL
  * > 15 years: 1.5 mg/dL
* Albumin >= 2 g/dL
* Female patients of childbearing potential must not be pregnant or breast-feeding; female patients of childbearing potential must have a negative serum or urine pregnancy test
* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study and for 6 months after the last drug administration
* Ability of subject or parent/guardian to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients with known inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy
* Only tumor types listed above are allowed; low grade gliomas (with and without neurofibromin 1 [NF1]) and ependymomas are excluded
* History of hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to murine protein-containing products
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with p28

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing dose-limiting toxicities (DLT) defined as any adverse event or grade 3 or 4 toxicity graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 6 weeks

SECONDARY OUTCOMES:
Percentage of patients whose tumors are p53 positive (greater than or equal to 10% of tumor cells staining for p53) | Up to 30 days post-treatment
  Will be estimated with its exact 95% confidence interval (CI).
Type and frequency of p53 mutations present in the tumor specimens analyzed | Up to 30 days post-treatment
  Will be summarized.
Change in tumor size | Baseline to up to 30 days post-treatment
  The proportion (and 95% CI) of subjects with an on-treatment tumor response or with clinical benefit will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - National Cancer Institute Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
As determined in the Clinical Trial Agreement